CLINICAL TRIAL: NCT06786091
Title: Late Side-effects After Cervical Cancer Treatment - Prevention and Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Sykehuset Ostfold (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 234097; 2023/FO426546 (Other Grant/Funding Number: Foundation Dam)
Record Dates: First submitted 2025-01-03; First posted 2025-01-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Floor Disorder; Female Pelvic Floor Dysfunction; Female Sexual Dysfunction; Female Urinary Incontinence; Fecal Incontinence; Secondary Lymphedema; Pelvic Pain
Keywords: feasibility studies; cervical cancer; pelvic floor muscle training; quality of life; pelvic floor morphology; pelvic floor muscle strength
MeSH Terms: conditions — Pelvic Floor Disorders; Fecal Incontinence; Pelvic Pain; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital pelvic floor exercise group (Experimental)
  Interventions: Other: Pelvic floor muscle training rehabilitation

INTERVENTIONS:
Other: Pelvic floor muscle training rehabilitation — The intervention consists of both exercise training, including pelvic floor muscle training, and information about the use of a dilator. At the baseline assessment participants are individually instructed in correct voluntary pelvic floor muscle contractions and how to perform intensive pelvic floor muscle training. The pelvic floor rehabilitation is supported with written information. The exercise program is provided with supervised digital group exercise sessions twice weekly and a home exercise program 4-5 weekly for 16 weeks. The home exercise program will be individualized if needed. The pelvic floor muscle training is following the recommendations for effective training dosage i.e. 3 sets of 10-12 repetitions, 5-7 times per week.

SUMMARY:
Late side-effects following gynecological cancer are predominantly symptoms from the pelvic region originating from the bowels, urinary tract, lymphatic system, genitals and musculoskeletal system. Pelvic floor dysfunctions such as urinary- and anal incontinence, pelvic organ prolapse, vaginal stenosis as well as compromised sexual function and dyspareunia appear to be highly prevalent. The incidence of gynecological cancer in Norway was 1700 in 2020 and the survival rate in Norway is among the highest in the world. Most women with cervical cancers are treated with curative intension and life expectancy at 5 years after diagnosis is >80%.

A negative impact of pelvic floor disorders on psychosocial well-being and quality of life are seen in survivors of gynecological cancer, and in cancer survivors this is found to be directly linked with patients regaining continence. Pelvic floor muscle training has few or no side effects, and is acknowledged as first line treatment for all types of urinary incontinence in women. Even though less studied, there is evidence to support pelvic floor muscle training as a safe intervention to reduce symptoms of anal incontinence and improve sexual function. A recent comparative cross-sectional study found that survivors of gynecological cancer with dyspareunia had higher stiffness and lower flexibility, coordination and endurance of the pelvic floor muscles compared to women with a history of total hysterectomy but no pelvic pain. These findings suggest a possible role for pelvic floor muscle training in the prevention and treatment of pelvic floor disorders after gynecological cancer. However, the overall quality of evidence for strengthening the pelvic floor muscles to reduce symptoms of pelvic floor dysfunctions after treatment of gynecological cancer is low.

This study aims to assess the feasibility of a digital pelvic floor rehabilitation programme led by an experienced pelvic floor physiotherapist. Study subjects are women treated for cervical cancer within the past 5 years, and all included participants will receive the intervention due to the feasibility design. Participants will be assessed clinically at baseline and endpoint, partly to ensure proper pelvic floor muscle contraction. The digital intervention ensures residents in rural areas equal access to specialized pelvic floor rehabilitation.

DETAILED DESCRIPTION:
Introduction:

The primary goal of cancer treatment is to cure the disease or considerably prolong life, and secondary to improve the patient's quality of life. However, more than 500 distinct kinds of late side effects have been associated with modern cancer therapy ranging from minor, asymptomatic changes to life-threatening injuries and death. Many cancer survivors do not regain their previous level of health and functioning. Thus, as life expectancy after cancer is increasing, more people are living with substantial and permanent bodily changes negatively affecting quality of life. Based on this, the Norwegian Women's Public Health Association (N.K.S.) has identified a knowledge gap in cancer treatment, with a main focus on prevention and treatment on late side-effects in "cancer affecting women" in the strategic research plan for 2018-2024.

Gynecological cancer includes cancer in the cervix, uterus, ovaries/fallopian tubes and vulva with an estimated global prevalence of 1.31 million new cases each year. Women diagnosed with uterine-, ovarian/fallopian tube and vulvar cancer are on average aged >60 years, while women diagnosed with cervical cancer are younger with a median age of 45 years. The incidence of gynecological cancer in Norway was 1700 in 2020b and the survival rate in Norway is among the highest in the world. Most women with cervical cancers are treated with curative intension and life expectancy at 5 years after diagnosis is >80%.

Late side-effects following gynecological cancer are predominantly symptoms from the pelvic region originating from the bowels, urinary tract, lymphatic system, genitals and musculoskeletal system. Pelvic floor dysfunctions such as urinary- and anal incontinence, pelvic organ prolapse, vaginal stenosis as well as compromised sexual function and dyspareunia appear to be highly prevalent. According to a recent systematic review including 31 studies of pelvic floor disorders in gynecological cancer survivors, prevalence of urinary incontinence was reported up to 76%, fecal incontinence up to 37% and dyspareunia up to 58%. However, study quality tended to be poor, and the need for more comparative data on pelvic floor disorders among gynecological cancer survivors and the general population is highlighted by several studies included in the review. A negative impact of pelvic floor disorders on psychosocial well-being and quality of life are seen in survivors of gynecological cancer, and in cancer survivors this is found to be directly linked with patients regaining continence.

Pelvic floor muscle training has few or no side effects, and is acknowledged as first line treatment for all types of urinary incontinence in women, and mild-moderate pelvic organ prolapse. Even though less studied, there is evidence to support pelvic floor muscle training as a safe intervention to reduce symptoms of anal incontinence and improve sexual function. The pelvic floor muscles is a three-layered muscle group covering the inside of the pelvis constituting the "floor" of the truncus. This muscle group encloses the urethra, vagina and rectum, and is involved in the continence mechanism, elimination, sexual arousal and support of the pelvic organs. There is evidence that structured pelvic floor muscle training increases muscle volume and stiffness, closes the levator hiatus and elevates the resting position of bladder and rectum.

Gynecologic cancer therapy often includes multiple treatment modalities, all which alone and in combination have the potential to affect the pelvic organs and the musculoskeletal system. Nonetheless, it is likely that pelvic floor disorders following cancer treatment are associated, at least in part, with a deterioration in pelvic floor muscle function. The functional properties of the pelvic floor muscles following treatment of gynecological cancer is poorly studied. One small study found that both passive and contractile properties of the pelvic floor muscles was altered in women with urinary incontinence following surgery and radiotherapy of stage I and II endometrial cancer compared to women with urinary incontinence after benign hysterectomy. A recent comparative cross-sectional study found that survivors of gynecological cancer with dyspareunia had higher stiffness and lower flexibility, coordination and endurance of the pelvic floor muscles compared to women with a history of total hysterectomy but no pelvic pain. These findings suggest a possible role for pelvic floor muscle training in the prevention and treatment of pelvic floor disorders after gynecological cancer.

Nevertheless, the overall quality of evidence for strengthening the pelvic floor muscles to reduce symptoms of pelvic floor dysfunctions after treatment of gynecological cancer is low. Some studies suggest a positive outcome of pelvic floor muscle training on symptoms of urinary incontinence, however these results lack statistical power and must be interpreted with caution. There is evidence to suggest that pelvic floor muscle training improves sexual function and dyspareunia, whereas there is scarce documentation of pelvic floor muscle training as treatment for anal incontinence following gynecological cancer. There is no clear evidence that regular vaginal dilatation reduces or prevent the risk of vaginal stenosis after pelvic radiotherapy. However, observational studies suggest a positive association with lower rates of self-reported stenosis, and recommending regular vaginal dilation after radiotherapy is established practice. Low compliance rates have been noted, and lack of sufficient information are the most commonly reported barrier, resulting in uncertainty about dilator use. Recently, Cyr et al. (2020) shoved good feasibility and acceptability of multimodal pelvic floor physical therapy, including pelvic floor muscle training and use of a dilator, for gynecological cancer survivors with dyspareunia. The intervention also led to significant improvements in pain, sexual function, pelvic floor dysfunction symptoms and quality of life.

Over the past decade there has been increasing research and clinical interest in the role of exercise as an adjunct therapy to improve symptom control and management following cancer diagnosis. More recently the research field has been extended beyond symptom control to also include evaluation of benefits for cancer-specific outcomes, cancer progression and metastasis. Overall, general exercise is recommended for cancer survivors and there is evidence that exercise may improve cancer-related health outcomes such as anxiety, symptoms of depression, body image/self-esteem, sleep disturbance, fatigue, physical functioning and health-related quality of life. Despite this, adherence to the recommended physical activity and exercise guidelines among cancer patients appears to be poor. A recent systematic scoping review found that cancer patients believed that physical activity and exercise was beneficial for their physical health and well-being. However, lack of support and treatment related side effects acted as barriers. Group exercising with other cancer patients who face similar challenges was a major facilitator among most participants. The authors calls for innovative healthcare products and technologies designed to help manage cancer related side effects and enhance compliance to physical activity and exercise guidelines.

The adverse effects from the pelvic region may have a slow trajectory of onset and are thus more prone to being overlooked by clinicians after the initial stages of treatment is over. Radical surgical interventions result in immediate symptoms with the potential for improvement with time, whereas radiation tends to elicit late effects that manifest over many months. As such, pelvic floor dysfunctions and sexual morbidity remains a neglected aspect of routine follow-up for cancer, and the user organization highlights the need for increased focus on sexual health in cancer rehabilitation. The topic is still a taboo inhibiting both patient and health care professionals, resulting in patients suffering with symptoms for a long time without seeking help. Community-based studies have shown that embarrassment, lack of knowledge about the causes, unfamiliarity with treatment options and the presence of concomitant symptoms are reasons for not seeking medical treatment. A qualitative study among gynecological cancer survivors found that most women reported their pelvic floor dysfunctions to be a direct consequence of the cancer treatment. Despite severe symptom burden and negative impact on quality of life, most women found their own ways of coping with these symptoms. Lack of knowledge about existing treatment options was the most frequently reported reason for not seeking help. In the same study, 11 out of 15 informants stated that post-treatment care should be improved with regards to information, prevention and management of pelvic floor disorder.

To summarize, surgery, radiotherapy and chemotherapy alone or in combination may induce detrimental long-term side-effects in survivors of gynecological cancer. In parallel, advances in cancer treatment improve survival rates and in combination with an increasingly older population, more women are living with adverse effects of cancer and cancer treatment. These developments have transformed the experience of cancer from a potentially life threatening illness, to the current interpretation of cancer as a long-term or chronic condition. Unfortunately, there is less focus on how to prevent late side-effects, and even less on how to treat them. This project aims to improve the knowledge base on prevention and treatment of late side-effects following gynecological cancer. More specific, the project objective are to assess:

Feasibility of a web-based education and exercise rehabilitation intervention to reduce late side-effects following treatment of cervical cancer.

Novelty and ambition:

The project is a response to research needs identified by the N.K.S. on "cancer affecting women" and "sexual and reproductive health". Further the project concurs with the N.K.S. research strategy 2018-2024 to reduce health discrepancies through equal access to healthcare. The project is according to Stiftelsen Dam's area of attention "patient and user centered research" aiming to promote health and quality of life and prevent known late effects in gynecological cancer survivors.

The novelty of this study is improving the knowledge of interventions preventing and reducing late side-effects of cervical cancer. The financial burden of late side-effects of cancer is large for patients as well as society. The financial burden may be further increased in the future with increasing direct costs related to medical care, and treatment for long-term side-effects, as well as indirect costs related to factors such as loss of productivity in combination with higher survival rates. Health literacy entails a person's knowledge, motivation and competences to access, understand, appraise and apply health information. During the life course, health literacy is vital and enables a person to evaluate and make informed decisions concerning health care, disease prevention and health promotion in order to maintain or improve quality of life. The Government's strategy (2020-2023)c aims to strengthen the active patient role with regards to health and treatment, and to facilitate services specifically tailored to the individual patient's needs. The use of new technology and health services that can be adapted to a greater extent in the patient's own home is highlighted.

The innovation potential in the present proposal is related to improved clinical pathways with increased focus on prevention and treatment of pelvic floor disorders. The intervention has a holistic approach with information and practical guidance empowering women to take on responsibility for their condition with appropriate clinical assessment, support and treatment. Exercise is a well-recognized and cost-effective intervention for musculoskeletal diseases in the general population, and results from this project will be the starting point of a full scale randomized controlled trial. Patient-centred care improves disease outcomes and quality of life and health literacy is mandatory for patients to make informed decisions and actions for themselves. A digitally supervised early education and rehabilitation intervention to prevent or reduce bothersome late side-effects following gynecological cancer will ensure patients equal access to specialized health care and rehabilitation regardless of where they live. Moreover, a digital intervention does not require physical attendance and is considered less burdensome as the patients do not need to travel and can follow the exercise group from their own homes. The intervention also facilitates contact with other survivors of gynecological cancer as the digital meetings opens 30 minutes prior to exercise to allow participants to chat with each other or ask questions to the physiotherapist. As the health care services are becoming more digitalized, the present proposal may also provide firsthand experience with digital exercise groups which may be useful to other clinical fields.

Research questions and hypotheses, theoretical approach and methodology:

The overall aim is to investigate the feasibility of an early digital education and exercise rehabilitation program.

Hypothesis:

A four month, twice weekly web-based education and exercise intervention is feasible and will result in a reduction in late symptoms of pelvic floor disorders and sexual dysfunction following treatment of cervical cancer.

Methodology:

The study design is an observational two-centre study. Participants and settings: Patients diagnosed with cervical cancer at St. Olavs Hospital, Trondheim University Hospital and Østfold Hospital Trust within the last five years are eligible for this study. We aim to include up to 40 women. Eligible women will be identified through outpatient cervical cancer control lists. We therefore apply exemption from the confidentiality principle. The unique eleven digit ID number will be used to invite eligible women through Eforsk. The inclusion criteria are women aged 18 years or over diagnosed and treated for cervical cancer (radical surgery or radiotherapy) within the last five years, cancer stadium I-III and adequate knowledge in Norwegian. Exclusion criteria are age >80 years, previous radiotherapy or pelvic surgery. Due to the design of a feasibility study, all included women will be offered the intervention. Study assessment visits: The clinical assessment visits are conducted with attendance at the outpatient clinic, Department of Physiotherapy. Baseline assessment will be done at study entry. Clinical assessment involves assessment of pelvic floor muscular strength and function. Strength and relaxation of the pelvic floor muscles are measured by a Camtech manometer. This involves the insertion of a small probe with a size smaller than a tampon into the vaginal opening. Further, strength and relaxation as well as muscular pain is assessed by internal palpation of the pelvic floor muscles in the vaginal opening. Some of the patients at St.Olavs hospital will be assessed by transperineal ultra sound imaging, involving an ultra sound probe at the perineum. The patients are reassessed after the 16-week intervention period. If the patient needs further individualized follow-up, contact will be established with a local primary health care physiotherapist. If relevant, patients will be referred to a gynecologist or sexual counselling.

Intervention:

The intervention consists of both exercise training, including pelvic floor muscle training, and information about the use of a dilator. At the baseline assessment participants are individually instructed in correct voluntary pelvic floor muscle contractions and how to perform intensive pelvic floor muscle training. The pelvic floor rehabilitation (pelvic floor muscle training and use of dilator) is supported with written information. The exercise program (aerobic and strength training, including pelvic floor muscle training) is provided with supervised digital group exercise sessions twice weekly and a home exercise program once weekly for 16 weeks. The home exercise program will be individualized if needed. The pelvic floor muscle training is following the recommendations for effective training dosage. The supervised digital exercise sessions are provided via www.join.nhn.no (Norsk Helsenett), and all sessions will open 30 minutes prior to exercise to allow for informal talk among participants and response to questions related to their treatment or training from the physiotherapist. Women will be offered individual video consultations for motivational talk in addition to the group sessions. Adherence to the exercise program is strongly emphasized and will be recorded in the patients' personal training diaries. Attendance in the digital group exercise will be registered by physiotherapists leading the group. Women not attending the group exercise sessions without prior notice will be contacted by telephone.

Outcome measures:

The primary outcome measures are to assess the willingness of participants to be included, their adherence and compliance to the intervention and response to the symptom questionnaires.

Secondary outcome measures are symptoms and severity of pelvic floor disorders, sexual function, lymphedema, quality of life and level of physical activity. Urinary incontinence are assessed using the International Consultation on Incontinence Questionnaire-UI Short Form (ICIQ-UI SF), an outcome measure developed to assess prevalence, severity, impact on quality of life and type of leakage. The short form has demonstrated satisfactory validity, reliability and sensitivity. Severity of anal incontinence symptoms is assessed with the widely used St.Marks incontinence score. The St. Marks score assesses frequency of stool and gas leakage, impact on daily life, urgency, pad use and use of constipating medication. Sexual dysfunction is assessed using the Amsterdam hyperactive pelvic floor scale (AHPFS) , the Female Sexual Distress Scale- revised (FSDS-R) and the Female Sexual Function Index. Quality of life is measured with The European Organization for Research and Treatment of Cancer Quality of Life core questionnaire (EORTC QLQ-C30) and QLQ-CX24. EORTC QLQ-C30 is a disease-specific instrument that is the instrument of choice in cancer trials in Europe. The EORTC QLQ-C30 incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and QOL scale. QLQ-CX24 is a cervical cancer-specific quality of life questionnaire module to be used in conjunction with QLQ-C30. Patient's impression of change is assessed by the Patient Global Impression of Change (PGIC). Secondary lymphedema will be assessed by the gynecologic cancer lymphedema questionnaire (GCLQ). Data regarding cancer diagnosis, treatment and potential medical events during the follow-up period will be collected from the patient medical records. Additionally, re-admission to hospital, ICD-10 diagnostic codes and in-hospital time will be recorded from the hospital records up to 12 months after completion of the chosen cancer treatment. In addition to the disease specific questionnaires, relevant baseline characteristics such as age, parity, type of delivery, menopause and vaginal supportive care, social status, education, frequency of physical activity, exercise activity and pelvic floor muscle training are collected on an digital questionnaire (eFORSK, https://www.klinforsk.no/info/Informasjon). Possible adverse events are recorded according to the CONSORT guidelines.

Statistics:

Statistical analysis include descriptive statistics, parametric tests for normal distributed data and non-parametric tests for skewed data

Sample size:

A power calculation is usually not advised when conduction a feasibility study, however, the sample size should be adequate to estimate critical parameters such as recruitment rate. Thus, it is suggested that recruiting 40 women may be sufficient.

User participation:

User involvement is ensured by including two members from patient interest organizations (Kreftforeningen and Gynkreftforeningen). The users are both survivors of gynecological cancer and trained in user involvement in research. So far, they have been consulted and provided valuable input on design of the intervention and follow-up. Further, they will be involved in the development and adaptation of the communication materials, and selection of questionnaires. The users are named as co-applicant for the funding and their time and travel expenses related to the project will be reimbursed. The phd-student will be the key person within the research team for users to contact. Further, N.K.S. research consultant Ida Heiaas and the N.K.S. "Womens health centre group" has contributed to the development of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed and treated for cervical cancer (surgery, radiation- or chemo therapy) within the last five years
* Cancer stadium I-III
* Adequate knowledge in Norwegian.

Exclusion Criteria:

- Previous pelvic radiation therapy or pelvic surgery.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility - participants willingness to be included | The time frame is pre-defined as one year recruitment period
  Participants willingness to be included (measured by inclusion rate i.e. how many are included out of the total number asked)
Adherence - participants adherence to the intervention | From enrollment until the end of the treatment at 16 weeks
  Participants adherence to the intervention, measured by how many group exercises they part-take in out of the total number of 32 group exercises
Compliance to home exercises | From enrollment until the end of the treatment at 16 weeks
  Participants compliance to the intervention. Participants are encouraged to do home exercises 3 times weekly (equals 48 exercise sessions over the intervention period). This is measured through reports in their training diary.
Participants impression of change | From enrollment until the end of the treatment at 16 weeks
  Participants impression of change following the intervention, measured by the Patient Global Impression of Change. Scale from 1-7, higher score indicating better outcome.

SECONDARY OUTCOMES:
Symptoms of urinary incontinence | From enrollment until the end of the treatment at 16 weeks
  Measured by the International Consultation on Incontinence Questionnaire-UI Short Form, ICIQ-UI SF. Scale from 0-21, higher scores indicating worse outcomes.
Symptoms and severity of anal incontinence | From enrollment until the end of the treatment at 16 weeks
  Measured by the St.Marks incontinence score. Scale from 0-24, higher scores indicating better worse outcomes.
Symptoms of bowel dysfunction | From enrollment until the end of the treatment at 16 weeks
  Measured with the Low Anterior Resection Syndrome Score - LARS Score. Scale from 0-42, higher scores indicating worse outcome.
Symptoms of sexual dysfunction | From enrollment until the end of the treatment at 16 weeks
  Measured by the Female Sexual Function Index. Scale ranging from 2-36, higher scores indicating better outcomes.
Pelvic pain symptoms | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  Pelvic pain symptoms, possibly due to an abnormally high-toned pelvic floor muscle measured by the 16-item Amsterdam Complex Pelvic Pain Symptom Scale (ACPPS-16). Scores range from 16-80, higher scores indicating worse outcomes.
Symptoms of sexual distress | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  Measured with the FSDS-R Female sexual distress scale - revised. Scores range from 0-42, higher scores indicate greater sexual distress (worse outcome).
Quality of life questionnaire (EORTC QLQ-C30) | From enrollment until the end of the treatment at 16 weeks
  Measured with The European Organization for Research and Treatment of Cancer Quality of Life core questionnaire (EORTC QLQ-C30) ,higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Quality of life QLQ-CX24 | From enrollment until the end of the treatment at 16 weeks
  Measured with The European Organization for Research and Treatment of Cancer Quality of Life core questionnaire QLQ-CX24.higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Symptoms of secondary lower limb lymphedema | From enrollment until the end of the treatment at 16 weeks
  Measured with the Gynecologic Cancer Lymphedema Questionnaire (GCLQ). Scores range from 0 to 20, higher scores indicating worse outcome.
Pelvic floor muscle strength (digital palpation) | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  Measured with the Oxford scale, scores ranging from 0-5, higher scores indicating higher level of muscle strength.
Pelvic floor muscle strength (pressure manometer) | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  Pelvic floor muscle strength measured on a pressure manometer, higher pressure indicating higher strength level (the Camtech Manometer).
Pelvic floor muscle resting tone | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  Measured with a pressure manometer (the Camtech Manometer). Lower sores associated with lower resting tone, higher scores indicating higher muscle resting tone.
Pain sensitization of the vestibulum | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  Measured by the Q tip test, measured at a dichotomous level; presence of pain: yes/no
Pelvic floor muscle morphology | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  Expressed at the change in the levator hiatal area (4D ultrasound) and distance between the symphysis and the puborectal muscle (2D ultrasound). Transperineal ultrasound imaging is planned for some of the included patients as part of the feasibility design.
Physical activity (frequency) | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  How often are you physically active? (By physically active we mean for instance walking, cross country skiing, cycling, swimming, running, or doing sports/exercise). Categorical (1) never, 2) less than once per week, 3) once per week, 4) 2-3 times per week, 5) every day)
Physical activity (intensity) | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  If you do physical activity once per week or more; how hard do you exercise? Categorical; 1) Easy, without sweating or shortness of breath, 2) So hard that I sweat and get out of breath, 3) So hard that I go all out.
Physical activity (how long) | From baseline clinical examination until endpoint clinical examination (after 16 weeks intervention)
  How long are you physically active each time? Categorical; 1) Less than 15 minutes, 2) 15-29 minutes, 3) 30-60 minutes, 4) More than 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Signe Nilssen Stafne, Study Chair — St. Olavs University Hospital
Locations (2):
- Norway (2):
  - St.Olavs University Hopsital, Trondheim, Trøndelag
  - Østfold Hospital, Fredrikstad, Østfold fylke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] Deutekom M, Dobben AC, Dijkgraaf MG, Terra MP, Stoker J, Bossuyt PM. Costs of outpatients with fecal incontinence. Scand J Gastroenterol. 2005 May;40(5):552-8. doi: 10.1080/00365520510012172. PMID 16036507
- [Background] Xu X, Menees SB, Zochowski MK, Fenner DE. Economic cost of fecal incontinence. Dis Colon Rectum. 2012 May;55(5):586-98. doi: 10.1097/DCR.0b013e31823dfd6d. PMID 22513438
- [Background] Bjerre Trent P, Falk RS, Staff AC, Jorde D, Eriksson AG. Translation and cross-cultural adaptation of the Gynecologic Cancer Lymphedema Questionnaire and the Lower Extremity Lymphedema Screening Questionnaire. Int J Gynecol Cancer. 2023 Feb 6;33(2):231-235. doi: 10.1136/ijgc-2022-003979. PMID 36600491
- [Background] Eidenberger M. Patient-Reported Outcome Measures With Secondary Lower Limb Lymphedemas: A Systematic Review. J Adv Pract Oncol. 2021 Mar;12(2):174-187. doi: 10.6004/jadpro.2021.12.2.5. Epub 2021 Mar 1. PMID 34109049
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Abrams D, Davidson M, Harrick J, Harcourt P, Zylinski M, Clancy J. Monitoring the change: current trends in outcome measure usage in physiotherapy. Man Ther. 2006 Feb;11(1):46-53. doi: 10.1016/j.math.2005.02.003. PMID 15886046
- [Background] Perrot S, Lanteri-Minet M. Patients' Global Impression of Change in the management of peripheral neuropathic pain: Clinical relevance and correlations in daily practice. Eur J Pain. 2019 Jul;23(6):1117-1128. doi: 10.1002/ejp.1378. Epub 2019 Mar 18. PMID 30793414
- [Background] Rampakakis E, Ste-Marie PA, Sampalis JS, Karellis A, Shir Y, Fitzcharles MA. Real-life assessment of the validity of patient global impression of change in fibromyalgia. RMD Open. 2015 Sep 14;1(1):e000146. doi: 10.1136/rmdopen-2015-000146. eCollection 2015. PMID 26535150
- [Background] Fayers P, Bottomley A; EORTC Quality of Life Group; Quality of Life Unit. Quality of life research within the EORTC-the EORTC QLQ-C30. European Organisation for Research and Treatment of Cancer. Eur J Cancer. 2002 Mar;38 Suppl 4:S125-33. doi: 10.1016/s0959-8049(01)00448-8. PMID 11858978
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] DeRogatis L, Pyke R, McCormack J, Hunter A, Harding G. Does the Female Sexual Distress Scale-Revised cover the feelings of women with HSDD? J Sex Med. 2011 Oct;8(10):2810-5. doi: 10.1111/j.1743-6109.2011.02385.x. Epub 2011 Jul 19. PMID 21771282
- [Background] Derogatis L, Clayton A, Lewis-D'Agostino D, Wunderlich G, Fu Y. Validation of the female sexual distress scale-revised for assessing distress in women with hypoactive sexual desire disorder. J Sex Med. 2008 Feb;5(2):357-64. doi: 10.1111/j.1743-6109.2007.00672.x. Epub 2007 Nov 27. PMID 18042215
- [Background] Derogatis LR, Rosen R, Leiblum S, Burnett A, Heiman J. The Female Sexual Distress Scale (FSDS): initial validation of a standardized scale for assessment of sexually related personal distress in women. J Sex Marital Ther. 2002 Jul-Sep;28(4):317-30. doi: 10.1080/00926230290001448. PMID 12082670
- [Background] Saga S, Stafne SN, Dons V, Bratlie I, Spetalen S, Hagemann CT. Amsterdam complex pelvic pain symptom scale with subscales: Based on a Norwegian translation, psychometric assessment and modification of the Amsterdam hyperactive pelvic floor scale. Acta Obstet Gynecol Scand. 2023 Oct;102(10):1409-1423. doi: 10.1111/aogs.14665. Epub 2023 Sep 7. PMID 37675780
- [Background] Hagen S, Glazener C, Sinclair L, Stark D, Bugge C. Psychometric properties of the pelvic organ prolapse symptom score. BJOG. 2009 Jan;116(1):25-31. doi: 10.1111/j.1471-0528.2008.01903.x. Epub 2008 Oct 8. PMID 18947342
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Bø KM, S;. Pelvic floor and exercise science. In: Bø KB, B; Mørkved, S; Van Kampen, M, editor. Evicence-based physical therapy for the pelvic floor Bridging science and clinical practice: Elsevier; 2015.
- [Background] Bø K, Hagen R, Kvarstein B, Jørgensen J, Larsen S, Burgio K. Pelvic floor muscle exercise for the treatment of female stress urinary incontinence: III. Effects of two different degrees of pelvic floor muscle exercises. Neurourol Urodyn. 1990;9(5):489-502
- [Background] Cyr MP, Dumoulin C, Bessette P, Pina A, Gotlieb WH, Lapointe-Milot K, Morin M. Characterizing Pelvic Floor Muscle Function and Morphometry in Survivors of Gynecological Cancer Who Have Dyspareunia: A Comparative Cross-Sectional Study. Phys Ther. 2021 Apr 4;101(4):pzab042. doi: 10.1093/ptj/pzab042. PMID 33522584
- [Background] Dietz HP. Pelvic Floor Ultrasound: A Review. Clin Obstet Gynecol. 2017 Mar;60(1):58-81. doi: 10.1097/GRF.0000000000000264. PMID 28005595
- [Background] Tennfjord MK, Engh ME, Bo K. An intra- and interrater reliability and agreement study of vaginal resting pressure, pelvic floor muscle strength, and muscular endurance using a manometer. Int Urogynecol J. 2017 Oct;28(10):1507-1514. doi: 10.1007/s00192-017-3290-y. Epub 2017 Mar 16. PMID 28299404
- [Background] Tritter JQ, Calnan M. Cancer as a chronic illness? Reconsidering categorization and exploring experience. Eur J Cancer Care (Engl). 2002 Sep;11(3):161-5. doi: 10.1046/j.1365-2354.2002.00345.x. PMID 12296831
- [Background] Hazewinkel MH, Sprangers MA, Taminiau-Bloem EF, van der Velden J, Burger MP, Roovers JP. Reasons for not seeking medical help for severe pelvic floor symptoms: a qualitative study in survivors of gynaecological cancer. BJOG. 2010 Jan;117(1):39-46. doi: 10.1111/j.1471-0528.2009.02411.x. PMID 19874292
- [Background] Teunissen D, van Weel C, Lagro-Janssen T. Urinary incontinence in older people living in the community: examining help-seeking behaviour. Br J Gen Pract. 2005 Oct;55(519):776-82. PMID 16212853
- [Background] Shaw C, Tansey R, Jackson C, Hyde C, Allan R. Barriers to help seeking in people with urinary symptoms. Fam Pract. 2001 Feb;18(1):48-52. doi: 10.1093/fampra/18.1.48. PMID 11145628
- [Background] Margalith I, Gillon G, Gordon D. Urinary incontinence in women under 65: quality of life, stress related to incontinence and patterns of seeking health care. Qual Life Res. 2004 Oct;13(8):1381-90. doi: 10.1023/B:QURE.0000040794.77438.cf. PMID 15503833
- [Background] Fakhrian K, Sauer T, Dinkel A, Klemm S, Schuster T, Molls M, Geinitz H. Chronic adverse events and quality of life after radiochemotherapy in anal cancer patients. A single institution experience and review of the literature. Strahlenther Onkol. 2013 Jun;189(6):486-94. doi: 10.1007/s00066-013-0314-5. Epub 2013 May 2. PMID 23636349
- [Background] Jensen NBK, Potter R, Kirchheiner K, Fokdal L, Lindegaard JC, Kirisits C, Mazeron R, Mahantshetty U, Jurgenliemk-Schulz IM, Segedin B, Hoskin P, Tanderup K; EMBRACE Collaborative Group. Bowel morbidity following radiochemotherapy and image-guided adaptive brachytherapy for cervical cancer: Physician- and patient reported outcome from the EMBRACE study. Radiother Oncol. 2018 Jun;127(3):431-439. doi: 10.1016/j.radonc.2018.05.016. Epub 2018 Jun 4. PMID 29880222
- [Background] Elshahat S, Treanor C, Donnelly M. Factors influencing physical activity participation among people living with or beyond cancer: a systematic scoping review. Int J Behav Nutr Phys Act. 2021 Apr 6;18(1):50. doi: 10.1186/s12966-021-01116-9. PMID 33823832
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Bonner C, Nattress K, Anderson C, Carter J, Milross C, Philp S, Juraskova I. Chore or priority? Barriers and facilitators affecting dilator use after pelvic radiotherapy for gynaecological cancer. Support Care Cancer. 2012 Oct;20(10):2305-13. doi: 10.1007/s00520-011-1337-z. Epub 2011 Dec 8. PMID 22160621
- [Background] Haddad NC, Soares Brollo LC, Pinho Oliveira MA, Bernardo-Filho M. Diagnostic Methods for Vaginal Stenosis and Compliance to Vaginal Dilator Use: A Systematic Review. J Sex Med. 2021 Mar;18(3):493-514. doi: 10.1016/j.jsxm.2020.12.013. Epub 2021 Jan 29. PMID 33526400
- [Background] Miles T, Johnson N. Vaginal dilator therapy for women receiving pelvic radiotherapy. Cochrane Database Syst Rev. 2014 Sep 8;2014(9):CD007291. doi: 10.1002/14651858.CD007291.pub3. PMID 25198150
- [Background] Brennen R, Lin KY, Denehy L, Frawley HC. The Effect of Pelvic Floor Muscle Interventions on Pelvic Floor Dysfunction After Gynecological Cancer Treatment: A Systematic Review. Phys Ther. 2020 Aug 12;100(8):1357-1371. doi: 10.1093/ptj/pzaa081. PMID 32367126
- [Background] Li J, Huang J, Zhang J, Li Y. A home-based, nurse-led health program for postoperative patients with early-stage cervical cancer: A randomized controlled trial. Eur J Oncol Nurs. 2016 Apr;21:174-80. doi: 10.1016/j.ejon.2015.09.009. Epub 2015 Oct 21. PMID 26482004
- [Background] Rutledge TL, Rogers R, Lee SJ, Muller CY. A pilot randomized control trial to evaluate pelvic floor muscle training for urinary incontinence among gynecologic cancer survivors. Gynecol Oncol. 2014 Jan;132(1):154-8. doi: 10.1016/j.ygyno.2013.10.024. Epub 2013 Oct 29. PMID 24183730
- [Background] Yang EJ, Lim JY, Rah UW, Kim YB. Effect of a pelvic floor muscle training program on gynecologic cancer survivors with pelvic floor dysfunction: a randomized controlled trial. Gynecol Oncol. 2012 Jun;125(3):705-11. doi: 10.1016/j.ygyno.2012.03.045. Epub 2012 Apr 1. PMID 22472463
- [Background] Cyr MP, Dumoulin C, Bessette P, Pina A, Gotlieb WH, Lapointe-Milot K, Mayrand MH, Morin M. Feasibility, acceptability and effects of multimodal pelvic floor physical therapy for gynecological cancer survivors suffering from painful sexual intercourse: A multicenter prospective interventional study. Gynecol Oncol. 2020 Dec;159(3):778-784. doi: 10.1016/j.ygyno.2020.09.001. Epub 2020 Oct 1. PMID 33010968
- [Background] Bernard S, Moffet H, Plante M, Ouellet MP, Leblond J, Dumoulin C. Pelvic-Floor Properties in Women Reporting Urinary Incontinence After Surgery and Radiotherapy for Endometrial Cancer. Phys Ther. 2017 Apr 1;97(4):438-448. doi: 10.1093/ptj/pzx012. PMID 28201796
- [Background] Hoff Braekken I, Majida M, Engh ME, Bo K. Morphological changes after pelvic floor muscle training measured by 3-dimensional ultrasonography: a randomized controlled trial. Obstet Gynecol. 2010 Feb;115(2 Pt 1):317-324. doi: 10.1097/AOG.0b013e3181cbd35f. PMID 20093905
- [Background] Ferreira CH, Dwyer PL, Davidson M, De Souza A, Ugarte JA, Frawley HC. Does pelvic floor muscle training improve female sexual function? A systematic review. Int Urogynecol J. 2015 Dec;26(12):1735-50. doi: 10.1007/s00192-015-2749-y. Epub 2015 Jun 14. PMID 26072126
- [Background] Hagen S, Stark D. Conservative prevention and management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD003882. doi: 10.1002/14651858.CD003882.pub4. PMID 22161382
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Gerharz EW, Mansson A, Hunt S, Skinner EC, Mansson W. Quality of life after cystectomy and urinary diversion: an evidence based analysis. J Urol. 2005 Nov;174(5):1729-36. doi: 10.1097/01.ju.0000176463.40530.05. PMID 16217273
- [Background] Porter MP, Penson DF. Health related quality of life after radical cystectomy and urinary diversion for bladder cancer: a systematic review and critical analysis of the literature. J Urol. 2005 Apr;173(4):1318-22. doi: 10.1097/01.ju.0000149080.82697.65. PMID 15758789
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Rutledge TL, Heckman SR, Qualls C, Muller CY, Rogers RG. Pelvic floor disorders and sexual function in gynecologic cancer survivors: a cohort study. Am J Obstet Gynecol. 2010 Nov;203(5):514.e1-7. doi: 10.1016/j.ajog.2010.08.004. Epub 2010 Sep 24. PMID 20869691
- [Background] Neron M, Bastide S, Tayrac R, Masia F, Ferrer C, Labaki M, Boileau L, Letouzey V, Huberlant S. Impact of gynecologic cancer on pelvic floor disorder symptoms and quality of life: an observational study. Sci Rep. 2019 Feb 19;9(1):2250. doi: 10.1038/s41598-019-38759-5. PMID 30783163
- [Background] Schofield C, Newton RU, Cohen PA, Galvao DA, McVeigh JA, Mohan GR, Tan J, Salfinger SG, Straker LM, Peddle-McIntyre CJ. Health-related quality of life and pelvic floor dysfunction in advanced-stage ovarian cancer survivors: associations with objective activity behaviors and physiological characteristics. Support Care Cancer. 2018 Jul;26(7):2239-2246. doi: 10.1007/s00520-018-4069-5. Epub 2018 Feb 1. PMID 29392481
- [Background] Lindgren A, Dunberger G, Enblom A. Experiences of incontinence and pelvic floor muscle training after gynaecologic cancer treatment. Support Care Cancer. 2017 Jan;25(1):157-166. doi: 10.1007/s00520-016-3394-9. Epub 2016 Sep 5. PMID 27596267
- [Background] Osann K, Hsieh S, Nelson EL, Monk BJ, Chase D, Cella D, Wenzel L. Factors associated with poor quality of life among cervical cancer survivors: implications for clinical care and clinical trials. Gynecol Oncol. 2014 Nov;135(2):266-72. doi: 10.1016/j.ygyno.2014.08.036. Epub 2014 Sep 3. PMID 25192629
- [Background] Ramaseshan AS, Felton J, Roque D, Rao G, Shipper AG, Sanses TVD. Pelvic floor disorders in women with gynecologic malignancies: a systematic review. Int Urogynecol J. 2018 Apr;29(4):459-476. doi: 10.1007/s00192-017-3467-4. Epub 2017 Sep 19. PMID 28929201
- [Background] Sekse RJT, Dunberger G, Olesen ML, Osterbye M, Seibaek L. Lived experiences and quality of life after gynaecological cancer-An integrative review. J Clin Nurs. 2019 May;28(9-10):1393-1421. doi: 10.1111/jocn.14721. Epub 2019 Jan 11. PMID 30461101
- [Background] Trotti A, Colevas AD, Setser A, Rusch V, Jaques D, Budach V, Langer C, Murphy B, Cumberlin R, Coleman CN, Rubin P. CTCAE v3.0: development of a comprehensive grading system for the adverse effects of cancer treatment. Semin Radiat Oncol. 2003 Jul;13(3):176-81. doi: 10.1016/S1053-4296(03)00031-6. PMID 12903007